CLINICAL TRIAL: NCT05587166
Title: Ultrasound-Guided Oblique Short-Axis Adductor Canal Block: Can the Oblique Approach Facilitate Perineural Catheter Insertion: A Randomized Controlled Trial
Brief Title: Ultrasound-Guided Oblique Short-Axis Adductor Canal Block.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Ahmed, MD, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MD-63-2021
Record Dates: First submitted 2022-06-30; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Adductor Canal Block

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The transverse short-axis group (Active Comparator)
  Interventions: Other: ultrasound guided adductor canal block
- The oblique short-axis group: (Experimental)
  Interventions: Other: ultrasound guided adductor canal block

INTERVENTIONS:
Other: ultrasound guided adductor canal block — ultrasound-guided adductor canal block using oblique short-axis for catheter insertion

SUMMARY:
The ideal pain management for knee surgery should provide excellent analgesia while minimizing opioid consumption and allowing early mobilization and rehabilitation.

The use of the continuous technique in ACB allows the delivery of a larger quantity of local anaesthetic into the adductor canal than in the single-shot technique.

The usual approach for ultrasound-guided ACB catheter insertion is through short-axis in-plane approach in which the ultrasound transducer is applied horizontally over the femoral artery and saphenous nerve. In this approach, the catheter is inserted through a 90-degree angulation with the nerve which might make the catheter insertion difficult.

In the new oblique position, the catheter will be inserted in a less than 90-degree angulation. This study speculates that decreasing the angle of catheter insertion will make catheter insertion easier and faster.

ELIGIBILITY:
Inclusion Criteria:

* adult patients more than 18 years
* ASA I-III
* scheduled for unilateral knee surgery under spinal anesthesia with an adductor canal perineural catheter planned for postoperative pain control

Exclusion Criteria:

* Patient who had an allergy to any drug used in the study
* Patients with neuropathy of any etiology in the affected extremity, hepatic or renal failure.
* pregnant females
* Patients who are unable to communicate with the investigators and hospital staff

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-15 (Estimated); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
catheter placement time (minutes) | starting from time of syringe removal from placement needle to time of complete threading of the catheter at 20-cm mark measured in minutes and over 20 minutes

IPD SHARING:
Plan to Share IPD: Undecided